CLINICAL TRIAL: NCT01335789
Title: Effect of Oxytocin on Stress Response in Marijuana-dependent Individuals
Brief Title: Effect of Oxytocin on Stress in Marijuana Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Associate Professor of Psychiatry, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20274
Record Dates: First submitted 2011-04-08; First posted 2011-04-14 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Marijuana Dependence
Keywords: marijuana; substance abuse; drug abuse; marijuana dependence; drug addiction
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (Active Comparator): intranasal administration
  Interventions: Drug: Oxytocin
- saline (Placebo Comparator): intranasal administration
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Oxytocin — 40 IUs
  Other Names: Pitocin
  Arms: Oxytocin
Drug: Saline — 40 IUs
  Arms: saline

SUMMARY:
The purpose of this study is to evaluate how people who frequently use marijuana respond to a stressful task, and if a medication (oxytocin) affects this response.

DETAILED DESCRIPTION:
Stress is commonly associated with drug craving and relapse in substance-dependent individuals. Several studies indicate that hypothalamic neuropeptides may mediate behavioral response to stress. For example, preclinical and clinical investigations have indicated that the neuropeptide oxytocin exerts anxiolytic effects in stress paradigms. Several studies have indicated that oxytocin promotes trust, social bonding, and calmness; however, little is known about the potential anxiolytic affects of oxytocin in marijuana-dependent individuals. A preclinical study investigating the effects and mechanism of lithium on cannabinoid withdrawal in rats had positive findings, with increasing oxytocin levels hypothesized to moderate this effect (Cui et al, 2001). Given the anxiolytic nature of oxytocin, it may have a therapeutic role in ameliorating the negative affect commonly observed prior to relapse in marijuana-dependent individuals, as well as the anxiety associated with marijuana withdrawal. This pilot protocol will provide important preliminary data on the effect of oxytocin on stress in marijuana-dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
* Subjects must meet DSM-IV criteria for current marijuana dependence (within the past three months). While individuals may also meet criteria for abuse of other substances, they must identify marijuana as their primary substance of abuse and must not meet criteria for dependence on any other substance (except nicotine) within the last 60 days.
* Subjects must consent to remain abstinent from all drugs of abuse (except nicotine and marijuana) for a three-day period immediately prior to the CTRC admission. Subjects must abstain from marijuana for 24 hours prior to testing. By restricting marijuana use as proposed, subjects should not be under the acute effects of marijuana, and also may be experiencing mild withdrawal symptoms, the measurement of which is one of the outcome variables being tested.
* Subjects must consent to random assignment.

Exclusion Criteria:

* Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
* Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect physiological/subjective responses.
* Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect hormonal/neuroendocrine status.
* Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with subjective measurements.
* Subjects with current major depressive disorder or post-traumatic stress disorder as these disorders are associated with characteristic changes in stress response.
* Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents that interfere with hormonal measurements within one month of test session.
* Subjects taking any psychotropic medications, including SRI's or other antidepressants, opiates or opiate antagonists because these may affect test response.
* Subjects with any acute illness or fever. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
* Subjects who are obese (³ 20% over ideal weight) as this may interfere with hormonal status.
* Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for three days prior to the stress task procedure.
* Subjects meeting DSM-IV criteria for substance dependence (other than nicotine or marijuana) within the past 60 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee McRae-Clark, Pharm.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between and March 2011 and August 2011 through community advertisements.
Period: Overall Study
Arm/Group | Oxytocin | Saline
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Saline | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (6.3) | 22.9 (7.1) | 23.3 (6.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Stress (as Measured by Cortisol)
Description: Salivary cortisol samples were collected via passive drool to provide empirical assessment of stress reactivity. Reported here is salivary cortisol level 5 minutes following Trier Social Stress Task exposure (approximately 60 minutes post study drug/placebo administration). Trier Social Stress Task is a psychosocial laboratory stress task in which subjects deliver a speech and perform a math problem in front of a stranger audience.
Time Frame: 5 minutes following Trier Social Stress Task completion
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Oxytocin | Saline
Number analyzed (Participants) | 8 | 8
nmol/L | 1.8 [1.5 to 2.2] | 2.1 [1.7 to 2.4]

2. Secondary Outcome: Craving (as Measured by the Marijuana Craving Questionnaire)
Description: The MCQ is intended to measure marijuana craving in adults. It measures symptoms on four subscales: expectancy, purposefulness, emotionality, and compulsivity. The scale rates individual items from 1-7 with a composite scoring range of 12-84 and possible subscale scoring range of 3-21. Reported here is MCQ composite score 5 minutes following Trier Social Stress Task exposure (approximately 60 minutes post study drug/placebo administration). Trier Social Stress Task is a psychosocial laboratory stress task in which subjects deliver a speech and perform a math problem in front of a stranger audience.
Time Frame: 5 minutes following Trier Social Stress Task completion
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oxytocin | Saline
Number analyzed (Participants) | 8 | 8
units on a scale | 41.1 [32.4 to 49.8] | 53.4 [44.7 to 62.1]

3. Primary Outcome: Stress (as Measured by Subjective Report)
Description: Subjective report of stress was measured using a 0-10 Likert Scale (0=not at all, 10=extremely). Reported here is subjective stress level 5 minutes following exposure to the Trier Social Stress Task (approximately 60 minutes post study drug/placebo administration). Trier Social Stress Task is a psychosocial laboratory stress task in which subjects deliver a speech and perform a math problem in front of a stranger audience.
Time Frame: 5 minutes following Trier Social Stress Task completion
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oxytocin | Saline
Number analyzed (Participants) | 8 | 8
units on a scale | 2.4 [0.2 to 4.6] | 3.0 [0.8 to 5.2]

ADVERSE EVENTS:
Arm/Group | Oxytocin | Saline
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=8) | Saline (N=8)
nasal irritation (General disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 2 (2)
irritability (Psychiatric disorders) | 1 (1) | 0 (0)
unpleasant taste in mouth (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size, non-treatment seeking sample, predominantly male sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes